CLINICAL TRIAL: NCT02980705
Title: A Randomized, Double-blind, Placebo-controlled Phase 2a Study to Evaluate the Efficacy and Safety of Tildrakizumab in Subjects With Active Ankylosing Spondylitis or Non-radiographic Axial Spondyloarthritis
Brief Title: Efficacy and Safety Study of SUNPG1622
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated-Sponsor's decision
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLR_16_22
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Active Ankylosing Spondylitis or Non-Radiographic Axial Spondyloarthritis
MeSH Terms: conditions — Non-Radiographic Axial Spondyloarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SUNPG1622 I (Experimental): SUNPG1622 I dose
  Interventions: Drug: SUNPG1622 I dose
- Placebo (Placebo Comparator): Placebo dose
  Interventions: Drug: Placebo dose

INTERVENTIONS:
Drug: SUNPG1622 I dose — Injection
  Arms: SUNPG1622 I
Drug: Placebo dose — Injection
  Arms: Placebo

SUMMARY:
This is a randomized, double-Blind, placebo-controlled Phase 2a study to evaluate the efficacy and safety of SUNPG1622.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed written consent
* Subject is ≥ 18 years of age at time of Screening
* Subject must be on a stable dose of NSAID for ≥ 2 weeks prior to initiation of investigational product
* Subject has a negative test for TB within 4 weeks before initiating IMP

Exclusion Criteria:

* Subjects with known diagnosis of fibromyalgia or complex regional pain syndromes
* Active uveitis or symptomatic inflammatory bowel disease requiring therapy at screening
* Radiographic evidence of total ankylosis of the spine
* Subject has a planned surgical intervention between Baseline and the Week 24 evaluation for a pre-treatment condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-09-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- SPARC Site 1, Middleburg Heights, Ohio, United States
- SPARC site 3, Budapest, Hungary
- SPARC site 3, Elblag, Poland
- SPARC site 2, A Coruña, Spain

REFERENCES:
- [Derived] Peters E, Chou RC, Rozzo SJ, Yao SL, Fructuoso FJG. A Randomized, Double-Blind, Placebo-Controlled Phase 2a Study of Tildrakizumab Efficacy and Safety in Patients With Active Ankylosing Spondylitis. J Clin Rheumatol. 2023 Aug 1;29(5):223-229. doi: 10.1097/RHU.0000000000001973. Epub 2023 May 10. PMID 37162744

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was planned that 90 subjects with active AS and 90 subjects with nr-axSpA would be enrolled to ensure completion of 180 subjects. One hundred and one subjects with active AS were actually enrolled and randomized and 82 subjects completed the study.
Period: Overall Study
Arm/Group | SUNPG1622 I | Placebo
Started | 50 | 51
Completed | 42 | 40
Not Completed | 8 | 11
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 6 | 9
Not completed — withdrew participation | 0 | 1
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SUNPG1622 I | Placebo | Total
Number analyzed (Participants) | 50 | 51 | 101
Age, Customized [Mean (Standard Deviation); unit: years]
  Age, mean years (SD) | 39.8 (9.18) | 39.1 (11.00) | 39.5 (10.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 39 | 38 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 48 | 51 | 99
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 48 | 50 | 98
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Assessment of SpondyloArthritis International Society 20 Response Rates
Description: Percentage of subjects who achieve improvement of ≥ 40% and absolute improvement of ≥ 20 units from baseline in a visual analog scale (0 [no disease activity]-100 [high disease activity]). The results for this endpoint is as per the Cochran-Mantel-Haenszel Analysis of ASAS20 Response Rates (Full Analysis Set).
Time Frame: Week 24
Population: Cochran-Mantel-Haenszel Analysis of ASAS20 Response Rates at Week 24 by Cohort (Full Analysis Set)
Measure: Number; unit: percentage of participants
Arm/Group | SUNPG1622 I | Placebo
Number analyzed (Participants) | 50 | 51
percentage of participants | 74.00 | 80.39

2. Secondary Outcome: Assessment of SpondyloArthritis International Society 20 Response Rates
Description: Percentage of subjects who achieve improvement of ≥ 40% and absolute improvement of ≥ 20 units from baseline in a visual analog scale (0 [no disease activity]-100 [high disease activity]). The following are the specific time points at which the outcome measure was assessed and for which data are presented : Week 1, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24.
Time Frame: Week 1, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
Population: ASAS20 Response Rates up to Week 24 by Cohort (Full Analysis Set)
Measure: Number; unit: percentage of participants
Arm/Group | SUNPG1622 I | Placebo
Number analyzed (Participants) | 50 | 51
percentage of participants
  Week 24 | 74.00 | 83.67
  Week 20 | 68.00 | 59.18
  Week 16 | 64.00 | 57.14
  Week 12 | 50.00 | 46.94
  Week 8 | 40.00 | 36.73
  Week 4 | 30.00 | 22.00
  Week 1 | 16.33 | 20.00

ADVERSE EVENTS:
Time Frame: Week 72
Description: It is the approximate duration over which adverse event data were collected.
  Analysis of adverse events was performed in 3 Parts:
  Part 1: SUNPG1622→Placebo; from Day 1 to Week 24 Part 2: Treatment follow-up (SUNPG16221 dose injection); from Week 24 to Week 52 Part 3: Washout period between Week 52 and Week 72. In Part 3 of the study, all subjects underwent IMP washout and no subjects received SUNPG1622.
Groups:
- Part 1: SUNPG1622 or Placebo: Group 1: SUNPG1622 or Placebo; From Baseline to Week 24.
  Safety results are provided per the following:
  Group 1: Subjects recieved either SUNPG1622 or Placebo
- Part 2: Treatment Follow-up (SUNPG16221 Dose Injection): Group 2: Treatment follow-up (SUNPG16221 dose injection); from Week 24 to Week 52.
  Safety results are provided per the following:
  Group 2: Subjects recieved SUNPG1622
- Part 3: Washout: Group 3: Washout period between Week 52 and Week 72.
  Safety results are provided per the following:
  Group 3: washout period
Arm/Group | Part 1: SUNPG1622 or Placebo | Part 2: Treatment Follow-up (SUNPG16221 Dose Injection) | Part 3: Washout
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/101 | 0/101
Serious Adverse Events (participants affected / at risk) | 0/101 | 1/101 | 3/101
Other Adverse Events (participants affected / at risk) | 12/101 | 13/101 | 0/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: SUNPG1622 or Placebo (N=101) | Part 2: Treatment Follow-up (SUNPG16221 Dose Injection) (N=101) | Part 3: Washout (N=101)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperplasia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: SUNPG1622 or Placebo (N=101) | Part 2: Treatment Follow-up (SUNPG16221 Dose Injection) (N=101) | Part 3: Washout (N=101)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hyperplasia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site joint erythema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Glucose tolerance impaired (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT02980705/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT02980705/SAP_002.pdf